CLINICAL TRIAL: NCT00172848
Title: Mastery, Social Support and Depression of Patients With Major Depression
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700303
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study was to discuss the relation of mastery, social support and depression in patients with depressive disorder. Cross-sectional quantitive study and purposive sampling method were designed. Data collection and analysis was conducted through structural questionnaires (including demographics, social support scale, mastery scale, CESD scale) at a medical center in Taipei. Results showed that patients with depression whose degree of depression was negative correlated with mastery and social support, and mastery was positive correlated with social support. Regression statistics results showed that mastery, social support, age, loss of jobs can predict degree of depression up to 60 percent. The mastery was strongest independent predictable factor to degree of depression, and had partial or total mediate effects to age, loss of jobs, financial condition, and social support. The result of this study suggested that clinically the care of patients with depression should focus on their confidence in mastery and provide strategies to promote their confidence in mastery, which can effectively reduce the degree of depression of those patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with depression

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult
Dates: Start 2004-10; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Chuan Hsiung, Ph.D, Study Chair — Department of Nursing, National Taiwan Umiversity
Locations (1):
- Ping-Chuan,Hsiung, Taipei, Taiwan